CLINICAL TRIAL: NCT07017439
Title: Investigating the Adjunctive Use of B3-agonist in the Early Post-Rezum Procedure Period: A Randomized Controlled Trial
Brief Title: Investigating the Adjunctive Use of Mirabegron in the Early Post-Rezum Procedure Period
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS26978
Record Dates: First submitted 2025-04-22; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostate Hypertrophy(BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Single blinded, placebo controlled, randomized trial. Two arms, one is the intervention arm which will receive mirabegron post rezum procedure while the control arm will receive a placebo pill with non-medicinal ingredients.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirabegron post procedure (Experimental): In this arm, patients will receive a 30 day prescription of mirabegron post-procedure.
  Interventions: Drug: Beta-3 agonists (Mirabegron/Myrbetriq)
- Placebo pill post rezum (Sham Comparator): Patients in this arm will be given the placebo pill following their procedure.
  Interventions: Other: Placebo group post rezum

INTERVENTIONS:
Drug: Beta-3 agonists (Mirabegron/Myrbetriq) — Patients in this arm will receive the medication in pill form following their procedure
  Arms: Mirabegron post procedure
Other: Placebo group post rezum — Patients in this arm will receive the placebo pill following their procedure.
  Arms: Placebo pill post rezum

SUMMARY:
The investigators propose conducting a randomized controlled trial at the Men's Health Clinic to evaluate whether patients who start and continue mirabegron postoperatively after undergoing Rezum therapy experience enhanced patient-reported outcomes, improved quality of life (QoL), and comparable rates of adverse events. There are no predicted adverse events of this study. There are no identified potential harms of this study.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a highly prevalent condition in men that can affect up to 80% of men by the age 80 1 . Minimally invasive surgical therapies (MISTs) are a growing area of research to provide adequate symptoms relief while avoiding potential adverse side effects. The Rezum 2 study was able to demonstrate significant improvement in symptom scores as well as uroflow parameters with preserved sexual function, and has become a valuable tool in a urologist's armamentarium for the management of LUTS/BPH. Despite the ultimate symptomatic relief from surgical management of BPH, the most common unwanted adverse event post treatment is early storage voiding symptoms (ie urgency, frequency, nocturia, urge incontinence) in 30-40% of patients 3 . Beta-3 agonists (e.g., Mirabegron) are commonly used to treat overactive bladder (OAB) symptoms, offering a more favorable side-effect profile compared to anticholinergic medications. One notable advantage of Beta-3 agonists, particularly in patients with benign prostatic hyperplasia (BPH) and lower urinary tract symptoms (LUTS), is the low risk of urinary retention 4,5 . In fact, urinary retention was not reported in initial phase III trials. The concurrent management of OAB symptoms during BPH surgery has been explored, including pharmacologic and intravesical options 3,6 . However, evidence supporting their use in patients who have undergone Rezum therapy remains limited. This single-blinded randomized controlled study is to be conducted at the Men's Health Clinic in Winnipeg, Manitoba. All eligible patients who are to undergo Rezum BPH/LUTS are to be included in the study. Patient meeting inclusion criteria and exclusion criteria (see below) will be randomized to either 1 month of B3-agonist or placebo pill. Inclusion criteria: age > 50, symptomatic LUTS with IPSS ≥ 10, prostate volume 30-80cc on any imaging modality, Qmax between 5 and 15ml/s with minimum voided volume of 125cc, frequency ≥ 8 voids/day. Exclusion criteria: PVR greater than 300ml, active UTI within past week, previous surgical intervention for BPH, documented urethral stricture disease, bladder stones, active malignancy, any confirmed or suspected neurologic disease, hypertension, known insensitivity to B3 agonist, current catheter dependence, currently taking anticholinergic, B3 agonist. Follow-up/data measurements will occur pre-procedure, immediately post procedure, 1 week, 2 weeks, and 4 weeks following procedure. At time of consultation pre-procedure, baseline symptom scores, uroflow parameters will be obtained. Symptom scores and any possible adverse events will again be measured at 1, 2 and 4 weeks. Additionally, at 4 weeks uroflow parameters are to be repeated. For this randomized controlled trial, a sample size of 44 was calculated to detect a mean difference of 3 in the OABSS score, which has been identified in prior literature as the minimal clinically significant difference. This calculation assumes a significance level of 5% and a power of 90%. Accounting for a projected crossover rate of 0% in the control arm and 12.5% in the experimental arm, the adjusted sample size increases to 58 participants.

ELIGIBILITY:
Inclusion Criteria:

* age >50, symptomatic LUTS with IPSS ≥ 10
* prostate volume 30-80cc on any imaging modality
* Qmax between 5 and 15ml/s with minimum voided volume of 125cc
* frequency ≥ 8 voids/day.

Exclusion Criteria:

* PVR greater than 300ml
* active UTI within past week
* previous surgical intervention for BPH
* documented urethral stricture disease
* bladder stones
* active malignancy
* any confirmed or suspected neurologic disease
* hypertension
* known insensitivity to B3 agonist
* current catheter dependence
* currently taking anticholinergic or B3 agonist.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in symptom scores | Symptom scores will be taken pre-op at time of consultation and at 1, 2 and 4 week follow-up
  Change in the following symptoms scores IPSS-QOL (higher scores indicate worser outcomes)
Change in symptom scores | Symptom scores will be taken pre-op at time of consultation and at 1, 2 and 4 week follow-up
  Change in OABSS symptom scores. (higher scores indicate worse outcomes)

SECONDARY OUTCOMES:
Rate of successful catheter removal | Will be measured at the scheduled trial of void either 1 week or 2 weeks post-op
  Rates of successful trial of voids(TOV) post-op will be captured. If the catheter is removed it is a succesful TOV, if it is not it is considered a failed TOV.
Adverse events | Possible adverse will be captured at time of consultation pre-op and at 1, 2 and 4 week follow-ups.
  Adverse events will be captured and recorded post-op.
rate of Qmax improvement | Uroflow parameters will be captured at time of consultation pre-op and the 4 week follow-up post-op.
  Uroflow parameter
rates of post void residual | Uroflow parameters will be captured at time of consultation pre-op and the 4 week follow-up post-op.
  Uroflow test
time to max flow | Uroflow parameters will be captured at time of consultation pre-op and the 4 week follow-up post-op.
  Uroflow test

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Rezūm Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology, 126, — https://journals.lww.com/tcmj/fulltext/2023/35040/treating_overactive_bladder_symptoms_after.5.aspx
- See also: Treating overactive bladder symptoms after transurethral prostatic surgery for benign prostatic hyperplasia - Which medication to choose? — https://journals.lww.com/tcmj/fulltext/2023/35040/treating_overactive_bladder_symptoms_after.5.aspx
- See also: A phase III, randomized, double-blind, parallel-group, placebo-controlled, multicentre study to assess the efficacy and safety of the β₃ adrenoceptor agonist, mirabegron, in patients with symptoms of overactive bladder. — https://doi-org.uml.idm.oclc.org/10.1016/j.urology.2013.02.077